CLINICAL TRIAL: NCT06332235
Title: A Randomized Open Label Phase-II Control Trial to Evaluate the Efficacy and Safety of Silodosin in the Treatment of Lower Urinary Tract Symptoms in Taiwanese Population.
Brief Title: Efficacy and Safety of Silodosin in the Treatment of Lower Urinary Tract Symptoms in Taiwanese Population.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-F(I)-20220023
Record Dates: First submitted 2023-04-09; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2023-04

CONDITIONS: Human Trichinellosis
MeSH Terms: conditions — Trichinellosis | interventions — silodosin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experiment group: 1. Subject ≥ 20 years of age
  2. Newly diagnosed of acute brain injury with Foley insertion with 5 days
  Interventions: Drug: Silodosin 8 mg

INTERVENTIONS:
Drug: Silodosin 8 mg — Dosing schedule: Oral, once daily
  Other Names: Conventional treatment

SUMMARY:
To evaluate the therapeutic effects and safety of silodosin in the patients of acute brain injury with lower urinary tract symptoms.

DETAILED DESCRIPTION:
I.Test drug

1. Name: Silodosin 8mg/capsule
2. Dosage form: capsule (Silodosin)
3. Dose(s): 8mg
4. Dosing schedule: Oral, once daily
5. Mechanism of action: Silodosin blocks the α1A-adrenergic receptors in the prostate gland and urethra, causing smooth muscle relaxation. Since the intraurethral pressure of the urethra is reduced, urine can pass more easily and the urinary symptoms are relieved.
6. Pharmacological category: α1A-adrenergic receptor blocker

II.The process of the experiment (brief describe) Eligible subjects will be randomized to a study medication according to the randomization schedule (a 1:1 randomization ratio). There are 2 groups in this study, with group A (treatment group, silodosin 8mg, once daily, 8-week duration) and group B (control group).

III. The primary endpoint is the rate of Foley removal. The secondary endpoints are the rate of urinary tract infection, residual urine amount and the rate of re-on Foley.

ELIGIBILITY:
Inclusion Criteria:

* Subject ≥ 20 years of age
* Newly diagnosed of acute brain injury with Foley insertion with 5 days

Exclusion Criteria:

* Subjects with already in use of α1A-adrenergic receptor blocker used
* Subjects with urethral trauma
* Subjects with a history of prostate, penile, testicular, bladder, or urethral cancer or has received pelvic radiation, systemic chemotherapy, or intravesical chemotherapy
* Expected survival days for brain injury less than 28 days
* Subjects with a history of renal dysfunction (elevated creatinine (>2.0 mg/dL))
* Subjects with severe liver impairment (Child-Pugh score≧10)
* Subjects with CYP3A4 inhibitors (ketoconazole、clarithromycin、itraconazole、ritonavir) used
* Subjects with pregnancy
* Subject who has been in an investigational drug study in the past 3 months
* Subjects who is considered as ineligible for participation in this clinical study by the principle investigator or the co-investigator's judgement.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed of acute brain injury with Foley insertion with 5 days
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment criteria Efficacy | 56 day
  Efficacy: the rate of Foley removal
Assessment criteria Safety | 56 day
  Silodosin-related adverse events

SECONDARY OUTCOMES:
Assessment criteria Efficacy | 56 day
  Efficacy: the rate of urinary tract infection

CONTACTS AND LOCATIONS:
Overall Officials: IRB, Study Chair — Affiliation
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Sanmin District, Taiwan